CLINICAL TRIAL: NCT07252765
Title: Nutritional Management of the Patient With Type 2 Diabetes at Nutritional Risk or With Malnutrition in Clinical Practice. STARLIGHT Study
Brief Title: Nutritional Management of the Patient With Type 2 Diabetes at Nutritional Risk or With Malnutrition in Clinical Practice
Acronym: STARLIGHT
Status: Recruiting | Type: Observational
Sponsor: Outcomes'10 (Network)
Collaborators: Nestlé Health Science Spain (Industry)
Responsible Party: Sponsor
Other Study IDs: NES-2024-252-DiabetPlus
Record Dates: First submitted 2025-09-10; First posted 2025-11-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Malnutrition; Malnourishment; Drug-Induced Diabetes
Keywords: Metabolic control; Disease - realted malnutrition; Diabetes-specific formula; T2D; Oral nutritional supplementation; Type 2 Diabetes Mellitus; Malnourishment; Malnutrition; Drug-induced diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with T2D or with drug-induced diabetes and malnutrition or at risk of it

SUMMARY:
The objective of this observational study is to characterize the patient profile and nutritional treatment patterns of individuals with type 2 diabetes (T2D) or drug-induced diabetes who present with malnutrition, or are at risk of it, and who are prescribed a diabetes-specific oral nutritional supplement (ONS) that is high in calories and protein and contains soluble fiber.

Participants will complete a series of questionnaires during visits 1 and 3.

DETAILED DESCRIPTION:
1. Background and Rationale This study focuses on patients with type 2 diabetes mellitus (T2D) who also present with malnutrition or are at risk of developing malnutrition. These conditions negatively affect clinical and functional outcomes, increasing the likelihood of complications and hospitalizations. The use of diabetes-specific oral nutritional supplements (ONS)-characterized by a high caloric and protein content and enriched with soluble fiber-may contribute to improving clinical status, nutritional parameters, and quality of life. Nevertheless, current evidence from real-world clinical practice remains limited and heterogeneous.
2. Primary Objective To characterize the clinical and nutritional profile, as well as the nutritional treatment patterns, of patients with T2D and malnutrition or at risk of malnutrition who are prescribed a diabetes-specific ONS.
3. Secondary Objectives

   To assess changes in glycemic and metabolic control.

   To evaluate the nutritional and functional impact of the ONS.

   To analyze healthcare resource utilization and associated costs.

   To estimate patient adherence, compliance, and satisfaction with the prescribed ONS.

   To assess quality-of-life outcomes over a 6-month follow-up period.
4. Exploratory Objective To explore changes in muscle mass using nutritional ultrasound.
5. Study Design

   Multicenter, prospective, real-world evidence (RWE) study.

   Conducted across 12 hospitals in Spain.

   Three scheduled visits: baseline (V1), 3-month follow-up (V2), and 6-month final visit (V3).
6. Study Population A total of 334 adult patients with T2D and either nutritional risk or malnutrition, all of whom are prescribed a diabetes-specific ONS.
7. Collected Variables

   Sociodemographic: age, sex, education level, etc.

   Clinical and anthropometric: weight, muscle mass, comorbidities.

   ONS-related: product name, dosage, duration, modifications, palatability.

   Nutritional requirements: daily caloric, protein, fat, and carbohydrate needs.

   Healthcare resource utilization: hospital admissions, emergency visits, specialist consultations, and diabetes medication adjustments.

   Metabolic profile: HbA1c, fasting glucose, lipid panel, albumin, total protein, hemoglobin, liver enzymes, eGFR, and CRP.

   Functional assessment: SARC-F scale, handgrip strength, bioelectrical impedance analysis (BIA), nutritional ultrasound, and Timed Up and Go test.

   Patient-reported outcomes: NutriQoL® quality-of-life questionnaire, satisfaction survey, treatment adherence questionnaire, and ONS palatability scale.
8. Data Management and Analysis Data will be managed by Outcomes'10 and analyzed using STATA v.14. Descriptive and comparative analyses will be conducted to address the primary and secondary objectives. All data will be reviewed and pseudonymized to ensure patient confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with type 2 diabetes (T2D) or drug-induced diabetes
* Patients at nutritional risk according to MUST or presenting malnutrition according to GLIM criteria.
* Patients requiring a diabetes-specific oral nutritional supplement (ONS) that is high-calorie, high-protein, and contains soluble fiber in real-world clinical practice, and who have been prescribed such a supplement within the previous 7 days.
* Patients able to provide informed consent and complete the study questionnaires.

Exclusion Criteria:

* Patients participating in other studies or clinical trials related to malnutrition, or who, in the investigator's opinion, may alter the course of the study.
* Patients currently receiving or expected to receive other types of nutritional interventions involving supplements (oral or otherwise) or non-conventional feeding methods (e.g., feeding tubes).
* Patients with a history of metabolic/endocrine diseases (other than diabetes) or any other condition causing liver or kidney failure, defined as ALT > 3x ULN or eGFR < 30 ml/min/1.73 m², and according to the investigator's judgment.
* Patients expected to undergo any surgical intervention or require hospitalization due to a condition unrelated to the study during the study period.
* Patients with other conditions that, in the investigator's opinion, may interfere with adherence to the intervention or with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with type 2 diabetes (T2D) or drug-induced diabetes, at nutritional risk according to MUST and/or presenting malnutrition according to GLIM criteria, who require a diabetes-specific oral nutritional supplement (ONS) that is high-calorie, high-protein, and contains soluble fiber, and who have been prescribed such an ONS in real-world clinical practice within the previous 7 days
Sampling Method: Non-Probability Sample
Enrollment: 334 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Descriptive of study population | Baseline visit (V1)
  Descriptive information of the population at V1

SECONDARY OUTCOMES:
Percentage change of blood test parameters | From enrollment to end of treatment at 24 weeks
  Changes in blood test measures will be compared
Percentage of patients with improvement in the nutritional status | From enrollment to end of treatment at 24 weeks
  Changes in GLIM or MUST classifications
Associated cost at 6-month follow-up | From enrollment to end of treatment at 24 weeks
  They will be estimated by multiplying the number of units used by their unit cost (derived from eSalud and Botplus databases). Unit: Number of events; euros (€)
Adherence with prescribed oral nutritional supplement (ONS) | From enrollment to end of treatment at 24 weeks
  Participants will be categorized as compliant (≥80% consumption) or non-compliant (<80%).
Change in functional status of participants over time | From enrollment to end of treatment at 24 weeks
  Changes between visits in SARC-F scale categories
Change in NutriQoL® quality-of-life score | From enrollment to end of treatment at 24 weeks
  Patients will be classified according to a quality-of-life category (excellent, good, acceptable, poor, very poor). Test total scoring values.
Patient satisfaction of the ONS product at 6 months | From enrollment to end of treatment at 24 weeks
  Responses to the satisfaction questionnaires will be summarized as number and percentage of participants selecting each category at V3.
Patient palatability of the ONS product at 6 months | From enrollment to end of treatment at 24 weeks
  Responses to the palatability questionnaires will be summarized as number and percentage of participants selecting each category at V3.
Health resource use | From enrollment to end of treatment at 24 weeks
  Frequencies of treatment changes, administration route, specialist consultations, and hospitalizations will be recorded and quantitative variables (treatment dose, treatment duration, number and days of hospitalization, consultations) will be summarized using mean ± SD.
Change in nutritional status | From enrollment to end of treatment at 24 weeks
  It will be estimated according to GLIM or MUST classification
Percentage change in BMI | From enrollment to end of treatment at 24 weeks
  Weight and height will be combined to report BMI in kg/m2
Maximum prehensile strenght value | From enrollment to end of treatment at 24 weeks
  Probe: handgrip test by using a hand dynamometer
30" chair test | From enrollment to end of treatment at 24 weeks
  Test: a patient will have to stand-up and sit-down as maximim number of times in 30", from a chair, with both arms crossed in the chest.
Impedancimetry values | From enrollment to end of treatment at 24 weeks
  Test: bioimpedance

OTHER OUTCOMES:
Nutritional status at molecular level | From enrollment to end of treatment at 24 weeks
  Test: nutritional (morphofunctional) ecography

CONTACTS AND LOCATIONS:
Locations (12):
- Spain (12):
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Juan Ramón Jiménez, Huelva, Huelva
  - Hospital UniversitarioDoctor Negrín, Las Palmas de Gran Canaria, Las Palmas
  - Hospital La Princesa, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Virgen de la Victoria, Málaga, Malaga
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla
  - Hospital Universitario Virgen de la Macarena, Seville, Sevilla
  - Hospital La Fe, Valencia, Valencia
  - Hospital General de Valencia, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No